CLINICAL TRIAL: NCT04082377
Title: Effects of Two Different Stepwise Lung Recruitment Maneuvers on Patient Hemodynamics During Anesthesia for Laproscopic Surgery
Brief Title: Effects of Two Different Stepwise Lung Recruitment Maneuvers on Patient Hemodynamics During Laproscopic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahmoud Mahmoud Othman, professor of Anesthesia and surgical ICU, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MD/19.06.188
Record Dates: First submitted 2019-09-05; First posted 2019-09-09 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Recruitment
MeSH Terms: interventions — Tidal Volume

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The management was carried out by a member of research team only aware of allocation group. The participants ,outcome assessor, surgeons and nursing staff will be totally blind of randomization schedule. All postoperative clinical staff handling patient care will be also unaware of the aim of the work.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recruitment maneuver with tidal volume (RM TV) (Experimental): RMs were conducted under volume controlled ventilation with initial settings of a limit of peak inspiratory pressure at 40cmH2O, TV at 6 mL/kg PBW ,RR at 7 breaths/min, PEEP at 5 cmH2O, and I:E ratio at1:1. The TV was then increased by steps of 4 mL/kg PBW until plateau airway pressure (Pplt) was 40 cmH2O, after which 3 breaths were allowed. Finally, the limit of peak inspiratory pressure, TV, RR, and I:E ratio were reset at values equal to those preceding the RM. The ventilation protocol could be changed at any time when concerned about patient safety.
  Interventions: Procedure: Recruitment maneuver with tidal volume (RM TV)
- Recruitment maneuver by PEEP (RM PEEP) (Active Comparator): The ventilation protocol consisted of volume controlled mechanical ventilation, FiO2 0.4, inspiratory-to-expiratory (I:E) ratio at 1:2, and respiratory rate (RR) set to normocapnia 5 cmH2O PEEP.
  RMs was conducted under pressure controlled ventilation so ventilation technique will be changed, pressure-control mode will be started and inspiratory time is increased to 50% (inspiratory: expiratory ratio will be set to 1:1). Peak airway inspiratory pressure (Ppeak) will be initially set to 20 cmH2O for three breaths, and then PEEP will be increased in steps from 5 to10 cmH2O for five breaths, from 10 to 15 cmH2O for seven breaths, from 15 to 20 cmH2O for ten breaths while Ppeak increased to 40 cmH2O and will be maintained for three more breaths. Following ARM, volume control will be re-established using Vt 6 mL/kg and step-wise reductions in PEEP from 20 to 15 cmH2O for three breaths,and then to 5 cmH2O until the end of recruitment maneuver.
  Interventions: Procedure: Recruitment maneuver by PEEP (RM PEEP)

INTERVENTIONS:
Procedure: Recruitment maneuver with tidal volume (RM TV) — The ventilation protocol consisted of volume controlled mechanical ventilation, FiO2 0.4, inspiratory-to-expiratory (I:E) ratio at 1:2, and respiratory rate (RR) set to normocapnia (end-tidal CO2 partial pressure between 35 and 40mmHg, TV 6 mL/kg PBW and 5 cmH2O PEEP.
  RMs were conducted under volume controlled ventilation with initial settings of a limit of peak inspiratory pressure at 40cmH2O, TV at 6 mL/kg PBW (PBW = 50.0+0.905*((height in cm)-152.4) for men, and = 45.5+0.905*((height in cm)-152.4) for women) Brower, et al. 1999, RR at 7 breaths/min, PEEP at5 cmH2O, and I:E ratio at1:1. The TV was then increased by steps of 4 mL/kg PBW until plateau airway pressure (Pplt) was 40 cmH2O, after which 3 breaths were allowed. Finally, the limit of peak inspiratory pressure, TV, RR, and I:E ratio were reset at values equal to those preceding the RM.
  Arms: Recruitment maneuver with tidal volume (RM TV)
Procedure: Recruitment maneuver by PEEP (RM PEEP) — The ventilation protocol consisted of volume controlled mechanical ventilation, FiO2 0.4, in RMs was conducted under pressure controlled ventilation so ventilation technique will be changed, pressure-control mode will be started and inspiratory time is increased to 50% (inspiratory: expiratory ratio will be set to 1:1). Peak airway inspiratory pressure (Ppeak) will be initially set to 20 cmH2O for three breaths, and then PEEP will be increased in steps from 5 to10 cmH2O for five breaths, from 10 to 15 cmH2O for seven breaths, from 15 to 20 cmH2O for ten breaths while Ppeak increased to 40 cmH2O and will be maintained for three more breaths. Following ARM, volume control will be re-established using Vt 6 mL/kg and step-wise reductions in PEEP from 20 to 15 cmH2O for three breaths,and then to 5 cmH2O until the end of recruitment maneuver
  Arms: Recruitment maneuver by PEEP (RM PEEP)

SUMMARY:
Pneumoperitoneum with CO2 insufflation during laparoscopic surgery elevates the intrathoracic pressure through the elevation of the diaphragm, which in turn decreases the lung compliance .Alveolar recruitment (AR) refers to the dynamic process of opening collapsed lung units by increasing transpulmonary pressure. It increases the area of ventilated lung parenchyma, thus improving gas exchange and arterial oxygenation .During lung recruitment, a transient increase in transpulmonary pressure induced by an intentional increase in airway pressures, results in an increase in intrathoracic pressure and a decrease in venous return, leading to a decrease in left ventricular end-diastolic areas and in stroke volume.

DETAILED DESCRIPTION:
Pneumoperitonium for laproscopic surgery usually result in decrease total respiratory compliance due to cranial shift of the diaphragm. Alveolar recuirtment is applied hopefully to minimize lung atlectasis and open collapsed alveoli to maintain arterial oxygenation. The anantomical proximity of lungs and heart within the chest means that any increase in intrathoracic pressure could have major effect on cardiovascular functions.Up to now, far too little attention has been paid to the decrease in left ventricular performance owing to fluctuation within the- chamber within chamber system-that preciptate stroke volume and cardiac output reduction during recruitment maneuvers.Up to our knowledge, the effect of ARM on patient heamodynamics is still unclear. in this study, we will compare two different recruitment maneuvers on patient haemodynamics during laproscopic surgery.Therefore this study is designed to investigate the effect of two individualized recruitment maneuvers during anethesia for laproscopic surgery to encourage best arterial oxygenation with the least haemodynamic compromise. Accordingly we assume that recruitment by incremental stepwise PEEP by 5cmH2o with pressure controlled ventilation may be associated with better stroke volume stability without haemodynamic alteration in comparison to incremental stepwise tidal volume by 4ml/kg during volume controlled ventilation.

* Pre-oxygenation for 5 minutes will be done in all patients and they will receive 0.02 mg/Kg midazolam, 1-2 μg/Kg fentanyl, 2-2.5 mg/kg Propofol slowly IV until loss of verbal contact. atracurium 0.5 mg/kg to facilitate proper placement of endotracheal tube. All patients will be mechanically ventilated using volume control mode (VC mode) with tidal volumes of 6 ml/ PBWT, with respiratory rate 12 breath per minute (bpm) and PEEP 5 cmH2O to keep end tidal Carbone dioxide (ETCO2) at 30-35 mmHg. Anaesthesia will be maintained in all patients using (1-1.5) minimum alveolar concentration (MAC) of Sevoflurane in O2/air mixture with FIO2 (0.4).Patients will be randomly assigned to one of two equal groups, according to computer-generated randomization sequence:
* group 1 (RM TV ): Recruitment maneuver with tidal volume .
* group 2 (RM PEEP): Recruitment maneuver with positive end expiratory pressure.

Group 1 (RM TV):

The ventilation protocol consisted of volume controlled mechanical ventilation, FiO2 0.4, inspiratory-to-expiratory (I:E) ratio at 1:2, and respiratory rate (RR) set to normocapnia (end-tidal CO2 partial pressure between 35 and 40mmHg, TV 6 mL/kg PBW and 5 cmH2O PEEP.

RMs were conducted under volume controlled ventilation with initial settings of a limit of peak inspiratory pressure at 40cmH2O, TV at 6 mL/kg PBW (PBW = 50.0+0.905*((height in cm)-152.4) for men, and = 45.5+0.905*((height in cm)-152.4) for women) , RR at 7 breaths/min, PEEP at5 cmH2O, and I:E ratio at1:1. The TV was then increased by steps of 4 mL/kg PBW until plateau airway pressure (Pplt) was 40 cmH2O, after which 3 breaths were allowed. Finally, the limit of peak inspiratory pressure, TV, RR, and I:E ratio were reset at values equal to those preceding the RM. The ventilation protocol could be changed at any time when concerned about patient safety.

Group 2 (RM PEEP):

The ventilation protocol consisted of volume controlled mechanical ventilation, FiO2 0.4, inspiratory-to-expiratory (I:E) ratio at 1:2, and respiratory rate (RR) set to normocapnia (end-tidal CO2 partial pressure between 35 and 40mmHg, TV 6 mL/kg PBW and 5 cmH2O PEEP.

RMs was conducted under pressure controlled ventilation so ventilation technique will be changed, pressure-control mode will be started and inspiratory time is increased to 50% (inspiratory: expiratory ratio will be set to 1:1). Peak airway inspiratory pressure (Ppeak) will be initially set to 20 cmH2O for three breaths, and then PEEP will be increased in steps from 5 to10 cmH2O for five breaths, from 10 to 15 cmH2O for seven breaths, from 15 to 20 cmH2O for ten breaths while Ppeak increased to 40 cmH2O and will be maintained for three more breaths. Following ARM, volume control will be re-established using Vt 6 mL/kg and step-wise reductions in PEEP from 20 to 15 cmH2O for three breaths,and then to 5 cmH2O until the end of recruitment maneuver.Monitoring:

Hemodynamic monitoring : stroke volume (SV), stroke volume variation (SVV), stroke volume index (SVI), cardiac output (COP), cardiac index (CI), systemic vascular resistance (SVR), systemic oxygen delivery (DO2) and oxygen delivery index (DO2I) will be measured by Cardiac output non-invasive monitor (ICONTM, OSYPKA medical cardiotronic GMBH, Elixir, Germany). Heart rate (HR), mean arterial blood pressure (MAP), and arterial oxygen saturation (Sao2) will be measured using HP monitor.

Respiratory monitoring : calculated lung compliance (dynamic compliance = TV / (peak airway pressure - PEEP)(static compliance = TV /(plateau pressure -PEEP) , peak airway pressure and plateau pressure, calculated alveolar dead space((1.135*(Paco2-Eco2)/(paco2-0.005)), driving pressure ( plateau pressure - PEEP) and Horowitz index ((Pao2 / Fio2)*100).

Basel hemodynamic variables will be obtained before endotrachial intubation (T0), Basel respiratory variables will be obtained just after endotracheal intubation(T0), Then allvariables will be obtained after endotrachial intubation (T1), after insuflation(T2), Intraopertive (T3a= at 1st hour intraopertive, T3b= at 2nd hour intraopertive, T3c= at 3rd hour intraopertive), after desuflation of the abdomen (T4), at end of surgery(T5). At each time point, the haemodynamic parameters will be recorded as follow: just before the alveolar recruitment maneuver (ARM), after 2 minutes of ARM, after 5 minutes of ARM.

Rescue strategies:

1. Intraoperative hypoxemia (Spo2< 92%): rescue will be primarily performed by ↑Fio2 by 0.1 till reach 100%.
2. Intraopertive hypotension (systolic blood pressure < 90 mmHg):

   * Abort ARM strategy if warranted.
   * Fluid administration ( 500 cc hydroxyethyl starch or 500 cc blood transfusion if indicated).
   * Noradrenaline infusion (0.1mg/kg/min) is the last resort. Postoperative follow up: hemodynamic variables will be monitored at arrival to post operative care unit (PACU) (P1), and after 2 hours (P2).Also chest x-ray to exclude postoperative complications like atlectasis or pneumothorax .

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients with American Society of Anesthesiologists (ASA) physical status I - II .
2. Both sexes.
3. laproscopic surgeries.

Exclusion Criteria :

1. Patients younger than 20 years.
2. body mass index (BMI) < 25 and > 35.
3. patients with major cardiovascular problems with ejection fraction < 40 %.
4. patients with chronic obstructive pulmonary diseases.
5. patients with major hepatic or renal dysfunction.

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Cardiac stroke volume | During intra-operative mechanical ventilation time
  Change in the stroke volume alteration by less than 10- 20% % during recruitment maneuver in anesthesia for laproscopic surgery.

SECONDARY OUTCOMES:
Dynamic lung compliance | During intra-operative mechanical ventilation time
  Change of dynamic lung compliance by more than 20% above basal.
Intraoperative oxygenation | During intra-operative mechanical ventilation time
  Change of intraoperative oxygenation with oxygen delivery index more than 550 ml/min/m2.
Horowitz ratio (Pao2/Fio2) | During intra-operative mechanical ventilation time
  Change of intraoperative oxygenation with Horowitz ratio more than 350.
Alveolar dead space ratio | During intra-operative mechanical ventilation time
  Change of the calculated alveolar dead space ratio (vd/vt) by less than 15%.
Mean arterial blood pressure | During intra-operative mechanical ventilation time
  Maintain mean blood pressure not less than 60 mmHg.
Pulmonary complications | During first 2 hours postoperative period
  Number of patients with postoperative pulmonary complications like atelectasis or pneumothorax.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud M Othman, MD, Principal Investigator — Faculty of medicine,Mansoura University
Locations (1):
- Urology and nephrology center, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No